

Analysis Plan 

# STATISTICAL ANALYSIS PLAN

#### **MVX0006**

A randomized, double-blind, placebo-controlled, parallel group study to evaluate the safety, tolerability and immunogenicity of the three doses of Group B Streptococcus vaccine (GBS-NN/NN2 with Alhydrogel®) in elderly participants aged 55 to 75

**AUTHOR:** 

VERSION NUMBER AND DATE: V1.0, 19APR2024

\\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\\BIOS\\MinervaX\\GBS-Document:

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP

Author: Version Number: 1.0

> Version Date: 19APR2024

Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

# STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan V1.0 (Dated 19APR2024) for Protocol MVX006.

| | Name | Signature | Date (DDMmmYYYY) |
|-----------|-----------------------|---------------------|------------------|
| Author: | | Refer to eSignature | |
| Position: | Statistical Scientist | | |
| Company: | IQVIA | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date (DDMmmYYYY) |
|---|---|---|---|
| Approved By: | | Refer to eSignature | |
| Position: | Medical Expert, VP Clinical | Development | |
| Company: | MinervaX | | |
| Approved By: | | | |
| Position: | | | |
| Company: | | | |
| Approved By: | | | |
| Position: | | | |
| Company: | | | |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\MinervaX\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

# **OUTPUT TEMPLATES SIGNATURE PAGE**

Output Templates V1.0 (Dated 19APR2024) for Protocol MVX006.

| | Name | Signature | Date (DDMmmYYYY) |
|-----------|-----------------------|---------------------|------------------|
| Author: | | Refer to eSignature | |
| Position: | Statistical Scientist | | |
| Company: | IQVIA | | |

Upon review of this document, the undersigned approves this version of the Output Templates, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date (DDMmmYYYY) |
|---|---|---|---|
| Approved By: | | Refer to eSignature | |
| Position: | Medical Expert, VP Clinical | Development | |
| Company: | MinervaX | | |
| Approved By: | | | |
| Position: | | | |
| Company: | | | |
| Approved By: | | | |
| Position: | | | |
| Company: | | | |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\MinervaX\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

# **MODIFICATION HISTORY**

| Unique<br>Identifier for<br>this Version | Date of the<br>Document<br>Version | Author | Significant Changes from<br>Previous Authorized Version |
|---|---|---|---|
| 1.0 | 19APR2024 | | Not Applicable – First Version |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\MinervaX\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

# TABLE OF CONTENTS

| 1.<br>2. | INTRODUCTION | | |
|---|---|---|---|
| 2.1. | Primary Objective | | 8 |
| 2.2. | Secondary Immunological Objectives | | |
| 2.3. | Secondary Safety Objectives | | |
| 2.4. | Exploratory Objectives | | 8 |
| 3. | STUDY ENDPOINTS | | 9 |
| 3.1. | Primary Endpoints | | 9 |
| 3.2. | Secondary Immunological Endpoints | | 9 |
| 3.3. | Secondary Safety Endpoints | | 9 |
| 3.4. | Exploratory Endpoints | | 10 |
| 4. | STUDY DESIGN | | 10 |
| 4.1. | General Description | | 10 |
| 4.2. | Schedule of Events | | 11 |
| 4.3. | Changes to Analysis from Protocol | | 11 |
| 5. | PLANNED ANALYSES | | 12 |
| 5.1. | Safety Review Group (SRG) | | 12 |
| 5.2. | Final Analysis | | 12 |
| 6. | ANALYSIS SETS | | 12 |
| 6.1. | Entered Analysis Set | | 12 |
| 6.2. | Enrolled Analysis Set | | 12 |
| Docur | ment: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp_ops\BIGNN_NN2\MVX0006\Biostatistics\Documentation\SA | | |
| Autho | or: | Version Number: | 1.0 |

Template No.: CS\_TP\_BS016 Revision 7

Effective Date: 01Nov2021

Reference: CS\_WI\_BS005



Analysis Plan 

| 6.3. | Safety Analysis Set | 12 |
|---|---|---|
| 6.4. | Immunogenicity Analysis Set | |
| 6.5. | Per-protocol Set | |
| 7. | GENERAL CONSIDERATIONS | 13 |
| 7.1. | Summary Statistics | 13 |
| 7.2. | Treatment Summarization | 13 |
| 7.3. | Precision | |
| <b>7.4.</b><br>7.4 | Reference Start Date and Study Day | |
| 7.5. | Baseline | 15 |
| 7.6. | Retests, Unscheduled Visits and Early Termination Data | 15 |
| 7.7. | Common Calculations | 15 |
| 7.8. | Software Version | 16 |
| 8. | STATISTICAL CONSIDERATIONS | 16 |
| 8.1. | Missing Data | 16 |
| 9. | OUTPUT PRESENTATIONS | |
| 10. | DISPOSITION AND WITHDRAWALS | |
| 11.<br>12. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS PROTOCOL DEVIATIONS | |
| 12.<br>13. | MEDICAL HISTORY | |
| 13.<br>14. | MEDICATIONS | |
| 1 <del>4</del> . | STUDY MEDICATION EXPOSURE | 18 |
| 16. | IMMUNOGENICITY ANALYSIS | |
| 17. | SAFETY OUTCOMES | |
| 17. | SAFETT OUTCOMES | 1) |
| 17.1. | Adverse Events | 19 |
| | .1.1. TEAEs Leading to Discontinuation of Study Medication or Withdrawal from Study | |
| 17. | .1.2. Serious Adverse Events | 21 |
| Docu | ment: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp_ops\BIOS\MinervaX\GBS-<br>NN_NN2\MVX0006\Biostatistics\Documentation\SAP | |


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

| 17.2. | Deaths | 21 |
|---|---|---|
| <b>17.3.</b> 17.3. | Safety Laboratory Evaluations 1. Laboratory Reference Ranges | 21 |
| 17.4. | Vital Signs | 22 |
| 17.5. | Physical Examination | 22 |
| | DATA NOT SUMMARIZED OR PRESENTEDENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS | |
| | & Times | |
| Spellin | g Format | 23 |
| Presen | tation of Treatment Groups | 23 |
| I istina | 37 | 2: |

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\MinervaX\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

#### 1. Introduction

This statistical analysis plan (SAP) describes the rules and conventions to be used in the presentation and analysis of immunogenicity and safety data for Protocol MVX0006. It describes the data to be summarized and analysed, including specifics of the statistical analyses to be performed.

This SAP is based on protocol version 3.0, dated 03May2023.

#### 2. STUDY OBJECTIVES

# 2.1. Primary Objective

The primary objective is to evaluate the safety and tolerability of the GBS-NN/NN2 vaccine for 4 weeks after each dose of vaccine.

# 2.2. Secondary Immunological Objectives

- To evaluate IgG antibody response to the GBS-NN/NN2 vaccine at Day 197 (principal immunological endpoint)
- To evaluate IgG antibody responses induced by the three vaccine doses, on a 0-, 1- and 6-month regimen, in older adult participants 4 weeks after each vaccination
- To assess whether pre-existing antibody levels affect the vaccine-induced antibody response.
- To evaluate the immune response up to 6 months following the third dose; to be reported in an addendum to the main CSR

# 2.3. Secondary Safety Objectives

To evaluate the long-term safety profile of the GBS-NN/NN2 vaccine between Day 57 (28 days post second injection) to Day 168 and 6 months following the third dose (safety endpoint); to be reported in an addendum to the main CSR.

# 2.4. Exploratory Objectives



NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 



### 3. STUDY ENDPOINTS

# 3.1. Primary Endpoints

- Safety and tolerability, as determined by the occurrence of adverse events (AEs) consisting of local and systemic reactogenicity, within 7 days after vaccination (Days 1 through 8 post each dose of investigational medicinal product (IMP)
- Unsolicited AEs, including AE of special interest (AESIs), medically attended AEs (MAAEs) and serious AEs (SAEs) within 28 days after each vaccination
- AESIs, MAAEs, adverse reactions (ARs)/serious adverse reactions (SARs) leading to withdrawal from study

# 3.2. Secondary Immunological Endpoints

- Geometric mean antibody concentration in μg/mL for antibodies to the four individual alpha-like proteins (Alps) (Alp 1, Alp 2/3, Rib and AlpC)
- Geometric mean fold increase in antibody concentration for antibodies to the four individual Alps (Alp 1, Alp 2/3, Rib and AlpC)
- Seroconversion rate (proportion of participants with a 4-fold increase above baseline pre dose concentration) at any timepoint post vaccination
- Proportion of participants achieving antibody concentrations for antibodies to the four individual Alps (Alp 1, Alp 2/3, Rib and AlpC) above specific thresholds at Days 29, 57, 169, and 197 (these thresholds will be 1, 2, 4 and 8 µg/mL

# 3.3. Secondary Safety Endpoints

- Proportion of participants with any SAE from Day 57 (28 days post 2<sup>nd</sup> injection) to Day 168 and 28 days after 3<sup>rd</sup> vaccination (Day 197) up to Day 365
- Proportion of participants with MAAEs, AESIs, ARs/SARs requiring a medical consultation, and/or leading to withdrawal from study from 28 days after 3<sup>rd</sup> vaccination (Day 197) up to Day 365

 $\label{local-plan} Document: $$ \ \c 2dnetvnasc01p-lan1.quintiles.net\cp_ops\BIOS\MinervaX\GBS-ret\colored{Constraints} $$$ 

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

| <b>3.4.</b> | Expl | loratory | Endi | oints |
|-------------|------|----------|------|-------|
| | - | / | | |

| • |
|---|
| • |
| • |

# 4. STUDY DESIGN

# 4.1. General Description

The purpose of this Phase 1 trial is to study the safety and immunogenicity of two dose levels, in an older adult population, with and without underlying medical conditions, to assess whether the GBS-NN/NN2 vaccine could potentially be effective in an older adult population and warrant further development in this population.

This is a Phase I, randomized, double-blind, placebo-controlled, parallel group study. Eligible participants will be randomized pre dose on Day 1, once all eligibility criteria have been verified. There will be two cohorts comprising 30 healthy older adult participants each and two cohorts comprising 15 obese and/or diabetic older adult participants each (see Figure 1):

- Cohort 1 (30 healthy older adult participants) will receive three injections, each consisting of 50 μg of GBS-NN and 50 μg of GBS-NN2 bound to aluminium hydroxide or placebo in a 4:1 ratio (investigational medicinal product [IMP]: placebo)
- Cohort 2 (30 healthy older adult participants) will receive three injections, each consisting of 125 μg of GBS-NN and 125 μg of GBS-NN2 bound to aluminium hydroxide or placebo in a 4:1 ratio (IMP: placebo)
- Cohort 3 (15 obese and/or diabetic older adult participants) will receive three injections, each consisting of 50 μg of GBS-NN and 50 μg of GBS-NN2 bound to aluminium hydroxide or placebo in a 4:1 ratio (IMP: placebo)
- Cohort 4 (15 obese and/or diabetic older adult participants) will receive three injections, each consisting of 125 μg of GBS-NN and 125 μg of GBS-NN2 or placebo bound to aluminium hydroxide in a 4:1 ratio (IMP: placebo)

Approximately 90 participants will be randomized in four cohorts.

Participants will be involved in the study for approximately one year including screening and safety follow-up. The start of the study is defined as Day 1 when participants are randomised. Eligible participants will be administered a dose of GBS-NN/NN2 or placebo on three occasions: the first dose will be administered on Day 1, followed by the second and third doses 4 and 24 weeks later, respectively.,

Progression from Cohort 1 to Cohort 2 and Cohort 3 will only occur after the available safety/tolerability data from all participants in Cohort 1 who completed Visit 3 (7 days post first dose) have been assessed by a Safety Review Group (SRG). The SRG will review the safety data from all participants who have completed Visit 3 in Cohort 2 and

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\MinervaX\GBS-

NN NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Title of the state



Analysis Plan 

Cohort 3 to determine if participants in Cohort 4 could receive the IMP.

During the study, participants will attend study visits as described in the Schedule of Activities (SoA) [Table 1 in Section 1.3 of the protocol], up to safety follow-up visit at month 12. Safety assessments will be performed, and immunogenicity blood samples will be collected at study visits according to the SoA.

Figure 1: Study Schema



GBS-NN/NN2: Group B Streptococcus vaccine containing the N-terminal domains of the Rib, Alpha C, Alpha 1 and Alpha 2/3 proteins.

#### 4.2. Schedule of Events

Schedule of events can be found in Section 1.3 of the protocol.

# 4.3. Changes to Analysis from Protocol

There are no changes to analyses from protocol.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\\BIOS\\MinervaX\\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

Effective Date: 01Nov2021

Copyright © 2009, 2010, 2012, 2016, 2018, 2019, 2021 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.



Analysis Plan 

#### 5. PLANNED ANALYSES

The following analyses will be performed for this study:

- Analyses for Safety Review Group (SRG) meetings by means of blinded data
- Final Analysis

# 5.1. Safety Review Group (SRG)

Reporting for the SRG is to be handled by IQVIA (project management, medical advisor) with input from the study clinic and is outside the scope of this document.

# 5.2. Final Analysis

All final, planned analyses identified in this SAP will be performed by IQVIA Biostatistics following Sponsor Authorization of this Statistical Analysis Plan, Database Lock, and Unblinding of Treatment.

### 6. ANALYSIS SETS

# **6.1.** Entered Analysis Set

The Entered Analysis Set will contain all participants who provide informed consent for this study. Participants in this analysis set will be used for disposition summary.

# **6.2.** Enrolled Analysis Set

The Enrolled Analysis Set will contain participants who have met all eligibility criteria.

# 6.3. Safety Analysis Set

The Safety Analysis Set will contain all participants randomly assigned to the study treatment and who receive at least one dose of the study drug (GBS-NN/NN2 or placebo). Participants will be classified according to treatment received. Participants in this analysis set will be used for demographic, and primary and secondary safety analyses.

# 6.4. Immunogenicity Analysis Set

The Immunogenicity Analysis Set will contain all participants from the Safety Analysis Set with at least one

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\MinervaX\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

scheduled post dose blood sample collected and analysed for immunogenicity (valid and non-missing value). Participants will be classified according to treatment received. Participants in this analysis set will be used for all immunological analyses.

### 6.5. Per-protocol Set

The Per-protocol Set will contain all participants who receive all three doses of the study vaccine and provide evaluable samples for analysis of the principal immunological endpoint without any protocol deviation that could lead to its exclusion.

The "principal" immunological analysis will also be performed on the Per-protocol Set if the number of participants in the Per-protocol set differs by more than 5% from the number of participants in the Safety Analysis Set.

#### 7. GENERAL CONSIDERATIONS

The safety and immunogenicity summaries, data listings as well as the statistical analysis of the immunogenicity variables will be the responsibility of the study biostatistician at IQVIA.

# 7.1. Summary Statistics

For qualitative variables, the population size (N for sample size and n for available data) and the percentage (of available data) for each class of the variable will be presented. Quantitative variables will be summarized using descriptive statistics, including N (with data available, n), mean, standard deviation (SD), coefficient of variation (CV%) as appropriate, median, minimum, and maximum values. Geometric mean will be included for immunogenicity variables, where applicable. Coefficient of variation will not be presented for change from baseline results.

The exact two-sided 95% CIs for a proportion within a treatment group will be calculated using the Clopper-Pearson exact method.

The geometric mean titres (GMTs) or geometric mean concentrations (GMCs) calculations will be performed by taking the anti-log of mean of the log10 titer transformation. Confidence interval for geometric means will be derived by raising 10 to the confidence interval associated with mean of log10 values i.e. CI of geometric mean =  $10^{\circ}$  (CI for the mean of the log10 values). All participants in the analysis set of interest with valid data will be considered. Subjects whose antibody titers/concentrations are below the cut-off of the assay will be given a value of half the cut-off for the purpose of GMT/GMC calculation (i.e., if the titer/concentration value is reported as "<X", X/2 will be used).

#### 7.2. Treatment Summarization

In general, data will be presented for each treatment group, with placebo participants from healthy older adult

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\MinervaX\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

cohorts (pooled together) and obese and/or diabetic older adult cohorts (pooled together) summarized separately. Data for all study participants combined will also be presented when appropriate. Data summary results will be presented for the following treatment groups as appropriate:

- Healthy Older Adult (HOA) Placebo (Pooled from Cohorts 1 and 2)
- HOA GBS-NN/NN2 50 μg
- HOA GBS-NN/NN2 125 μg
- Obese and/or diabetic Older Adult (O/DOA) Placebo (pooled from Cohorts 3 and 4)
- O/DOA GBS-NN/NN2 50 μg
- O/DOA GBS-NN/NN2 125 μg
- All participants combined, if appropriate

#### 7.3. Precision

Quantitative safety data (clinical laboratory values, vital signs) and immunogenicity data will be reported to the same precision as the source data.

For the reporting of descriptive statistics, the mean, median, standard deviation, and confidence intervals will be presented to one digit more precision than the source data. The minimum and maximum will be presented to the same precision as the source data except for the below precision rules for geometric mean titers (GMT) or concentrations (GMC). Coefficient of variation (%) will always be reported to 1 decimal place. P-values, if any, shall be reported to four decimal places or as <0.0001.

The number of decimals used when displaying GMT or (Geometric Mean Concentrations (GMC) and their confidence limits is shown in the following table:

| GMT or GMC Value | Number of decimals to display |
|------------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMT/GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the one with the higher number of decimals). Geometric mean fold ratios (GMFRs) or GMT/GMC ratios and their confidence limits will be displayed with 1 decimal regardless of the actual values.

# 7.4. Reference Start Date and Study Day

Study Day will be calculated from the reference start date and will be used to show start/stop day of assessments and

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\MinervaX\GBS-

NN NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

events. Study day will appear in every listing where an assessment date or event date appears. Reference start date is defined as the day of the first dose of study medication (Day 1 is the day of the first dose of study medication).

- If the date of the event is on or after the reference date, then: Study Day = (date of event reference date) + 1.
- If the date of the event is prior to the reference date, then: Study Day = (date of event reference date).

In the situation where the event date is partial or missing, Study Day, and any corresponding durations will appear partial or missing in the listings.

#### 7.4.1. Attributing Events to Vaccine Doses

The dose relative to an event is the most recent study dose given to a subject prior to the start of a given event. For example, if the start date of an AE is between Dose 1 and Dose 2, the relative dose will be Dose 1.

#### 7.5. Baseline

Baseline is defined as the last scheduled non-missing measurement taken prior to dosing and will correspond to Day 1 pre-dose for immunogenicity assessments, clinical laboratory evaluations and vital signs. However, if a subject is missing the planned baseline collection, the previous non-missing scheduled evaluation will become the baseline value.

# 7.6. Retests, Unscheduled Visits and Early Termination Data

Unscheduled measurements will not be included in summary statistics. Early termination results will be recorded as such and included with the end-of-study summaries.

Listings will include all scheduled, unscheduled, retest and early discontinuation data.

#### 7.7. Common Calculations

For quantitative safety measurements (e.g., vital signs, laboratory evaluations), change from baseline will be calculated as:

• Test Value (after baseline) – Baseline Value

For immunogenicity measurements, fold change from baseline will be calculated as:

• Test Value (after baseline) / Baseline Value

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\MinervaX\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

#### 7.8. Software Version

All derivations, statistical analyses, summaries and listings will be generated using SAS version 9.4 or higher (SAS Institute, Inc., Cary, North Carolina).

#### 8. STATISTICAL CONSIDERATIONS

### 8.1. Missing Data

Missing safety data will not be imputed.

#### 9. OUTPUT PRESENTATIONS

Appendix 1 shows conventions for presentation of data in outputs.

The templates provided with this SAP describe the presentations for this study and therefore the format and content of the summary tables, figures, and listings to be provided by IQVIA Biostatistics.

Some minor modifications may be necessary to the planned design of tables, figures, and listings to accommodate data collected during the actual study conduct.

#### 10. DISPOSITION AND WITHDRAWALS

All subjects who provide informed consent will be accounted for in this study. Subject disposition will be tabulated for each study treatment and for all subjects combined with the number of subjects who are screened, eligible to be randomized, randomly assigned to treatment, complete the study, prematurely discontinue, and the reason for early discontinuation. A listing will present dates of completion or early withdrawal and the reason for early discontinuation, if applicable, for each subject.

Listings of study protocol deviations, study eligibility, treatment randomization, and study treatment administration will be provided.

# 11. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Individual subject demographics and baseline characteristics (medical history and serology screening) will be presented in listings.

Demographic characteristics such as age, sex, race, ethnicity, height, weight, and body mass index (BMI) will be summarized and tabulated by treatment and for all subjects combined. Descriptive statistics will be presented for

 $\label{local-pos} Document: $$ \c 2dnetvnasc01p-lan1.quintiles.net\cp_ops\BIOS\MinervaX\GBS-relation = $$ \c 2dnetvnasc01p-lan1.quintiles.net\c 2dnetvnasc01p-lan1.quintiles.net\c$ 

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

age, height, weight, and BMI. Frequency counts and percentages will be presented for sex, race, and ethnicity. No statistical testing will be carried out for demographic or other baseline characteristics.

#### 12. PROTOCOL DEVIATIONS

A deviation from a protocol occurs when Investigator site staff or a study participant does not adhere to the protocol's stipulated requirements, whether inadvertently or planned. Protocol deviations will be listed and will include a classification of critical, minor or major, as determined by Sponsor

Changes to the procedures or events, which may impact the quality of the immunogenicity data, will be considered important/significant protocol deviations and will be described within the clinical study report body text. These changes or events will include any circumstances that will alter the evaluation of the immunogenicity results. Examples include, but may not be limited to, sample processing errors that lead to inaccurate immunogenicity results, and/or inaccurate dosing.

In the case of a important/significant protocol deviation or event, immunogenicity data collected during the affected timepoint will be excluded from the immunogenicity analysis. Other changes to the procedures or events which do not impact the quality of the immunogenicity data will not be considered significant protocol deviations. A common example of a non-significant protocol deviation is a missed blood sample or deviations from blood collection times.

#### 13. MEDICAL HISTORY

Medical history coded using Medical Dictionary for Regulatory Activities (MedDRA) Version 26 or higher will be listed for the safety analysis set.

#### 14. MEDICATIONS

Medication usage will be coded using the WHO Drug Dictionary March 2022 or higher will be presented for the safety analysis set.

- 'Prior' medications are medications which started and stopped prior to the first dose of study medication.
- 'Concomitant' medications are medications which were taken during the treatment period, or specifically:
  - o started on or after the first dose of study medication or
  - started prior to the first dose of study medication and were continued after the first dose of study medication

Concomitant medications will be summarized using WHO Drug Class and preferred drug name.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\MinervaX\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

#### STUDY MEDICATION EXPOSURE 15.

Exposure to study medication, as the number of doses administered, will be presented for each treatment group in the Safety Analysis Set.

#### 16. IMMUNOGENICITY ANALYSIS

Listings of blood sample collection date and time for antibody and cellular response will be presented separately for participants within each treatment group. Individual observed values for secondary endpoints will be listed and summarized using descriptive statistics by treatment groups across all scheduled timepoints during the entire study.

The secondary immunogenicity endpoints are antibodies to the four individual Alps:

- Alp1 antibody concentration in µg/mL
- Alp2/3 antibody concentration in μg/mL
- Rib antibody concentration in µg/mL
- AlpC antibody concentration in µg/mL

For each treatment group, at each timepoint that samples are collected for antibody:

- GMCs and their 95% CI will be tabulated (GMC at Day 197 is the "principal" immunological endpoint)
- Geometric mean fold change from baseline with their 95% CI will be tabulated
- Proportion of participants with 4-fold increase from baseline (seroconversion)
- Proportion of participants with antibody concentrations above specific thresholds (1, 2, 4 and 8 µg/mL)

Linear mixed model with repeated measures (MMRM) will be used to perform pairwise comparison of the secondary endpoints between treatment groups separately for healthy older adults and obese/diabetic older adults. Results from Days 1, 29, 57, 169 and 197 will be utilized. The model will use fixed effects for treatment, day (as a categorical variable), treatment×day, and baseline value as a covariate, and a repeated day effect within a subject under an unstructured covariance matrix. Concentration values (i.e., the response variable) will be log10transformed prior to the analyses and then back-transformed for presentation. Least-squares adjusted GMC with associated 95% CI for individual treatments and adjusted geometric mean ratio, 95% CI and p-values for pairwise comparison will be presented from the fitted model. Variance between the treatment groups will not be considered equal. Age and sex will be included in the model as covariates. If unstructured covariance matrix leads to model convergence failure, then compound symmetric or auto-regressive AR(1) matrix will be tried in the order mentioned.

Analyses of exploratory endpoints are outside the scope of this plan and will be reported separately from the clinical study report.

Comparative analyses with placebo will be exploratory and should be interpreted with caution considering that there is no adjustment for multiplicity and that treatment group sizes are small for these comparisons. The immunogenicity analysis will be carried out on the immunogenicity analysis set. The "principal" immunological analysis will also be performed on the Per-protocol Set if the number of participants in the Per-protocol set differs

\\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\MinervaX\GBS-Document:

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

by more than 5% from the number of participants in the Safety Analysis Set.

The following figures will be produced for the antibody response (secondary endpoints) separately:

- Boxplots of the log10(concentration) per timepoint, stratified by treatment and healthy and obese/diabetic
- Boxplots of the fold-rise from baseline per timepoint, stratified by treatment and healthy and obese/diabetic
- Plots of the LS-adjusted GMCs over time with 95% CIs, stratified by treatment and healthy and obese/diabetic

# 17. SAFETY OUTCOMES

All outputs for safety outcomes will be based on the Safety Analysis Set.

There will be no statistical comparisons between the treatment groups for safety data, unless otherwise specified within the relevant section.

#### 17.1. Adverse Events

Adverse Events (AEs) will be coded using MedDRA central coding dictionary, Version 26 or higher.

Treatment emergent adverse events (TEAEs) are defined as AEs that started or worsened in severity on or after the first dose of study medication.

The number and percentage of participants with at least 1 solicited AE (local, systemic and any) during the 7-day solicited period will be tabulated by treatment group with exact 95% CI after each vaccination and overall.

The number and percentage of participants reporting individual solicited local and systemic AE during the 7-day solicited follow-up period will be tabulated by treatment group and severity grade with exact 95% CI as follows:

- Over the 3 doses, the percentage of subjects with the symptom and its exact 95% CI
- At each study dose (visit), the percentage of subjects with the symptom and its exact 95% CI

Counting rules for occurrences of solicited adverse events: When the occurrences of solicited adverse events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurred. For a given participant and the analysis of solicited symptoms within 7 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore, the analysis of the solicited AEs includes only vaccinated subjects for doses with documented safety data (i.e., ediary completed). More specifically the following rules will be used:

- Participants who documented the absence of a solicited symptom after one dose will be considered not having that symptom after that dose.
- Subjects who documented the presence of a solicited symptom and fully or partially recorded daily
  measurement over the solicited period will be included in the summaries at that dose and classified
  according to their maximum observed daily recording over the solicited period
- Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be assigned to the lowest intensity category at that dose (i.e. 38°C for fever or

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\MinervaX\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS TP BS016 Revision 7 Reference: CS WI BS005



Analysis Plan 

grade 1 for other symptoms)

• Doses without ediary completed will be excluded

The number and percentage of participants with unsolicited AEs within 28 days after any doses with its exact 95% CI will be tabulated by system organ class and preferred term for each treatment group. Similar tabulation will be done for

- severe (grade 3) unsolicited AEs
- unsolicited AEs causally related to vaccination
- severe and causally related unsolicited AEs
- unsolicited AEs of special interest (AESIs)
- unsolicited AEs requiring medical attendance (MAAEs)

The incidence of solicited adverse events (local and systemic) with severity will be plotted using horizontal bar charts. For the purpose of this plot, severity will follow the definitions according to the <u>FDA Guidance for Industry:</u> <u>Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (September 2007)</u>. For example, the result collected in eCRF will correspond to following severity grades:

#### Injection Site Pain:

Awareness of injection site pain, but easily tolerated: Mild or Grade 1
Injection site pain is affecting normal activities: Moderate or Grade 2

Unable to do normal activities, health is affected, and needs medication or visit: Severe or Grade 3

Systemic Events (Chills, Muscle Pains, Fatigue, Headache, Malaise, Nausea, Vomiting):

Awareness but easily tolerated: Mild or Grade 1 Affecting normal activities: Moderate or Grade 2 Unable to do normal activities: Severe or Grade 3.

# 17.1.1. TEAEs Leading to Discontinuation of Study Medication or Withdrawal from Study

Treatment emergent adverse events (TEAEs) leading to permanent discontinuation of study medication will be identified by using the variable "Action taken with study treatment" = "Permanently withdrawn" from the AE page of eCRF and will be listed.

TEAEs leading to withdrawal from study will be identified by using the variable "Did the subject withdraw from study due to this event" = "Yes" from the AE page of eCRF and will be listed.

The number and percentage of participants with AESIs, MAAEs, AEs/SAEs, and ARs/SARs leading to withdrawal from the study or discontinuation of the treatment will be tabulated by SOC and PT.

The number and percentage of participants with any SAE, AESIs, MAAEs, ARs/SARs leading to withdrawal from the study between Day 57 (28 days post second injection) to Day 168 and from 28 days after third vaccination up to Day 365 will be summarised by treatment group and by SOC and PT.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\MinervaX\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

Note: Adverse reactions (ARs) are defined as adverse events considered related to vaccination.

#### 17.1.2. **Serious Adverse Events**

Participants who experienced at least 1 SAE within 28 days after any dose, from dose 1 until 28 days post last dose and during the entire study period will be listed.

The number and percentage of participants with any SAE and SARs between Day 57 (28 days post second injection) to Day 168 and from 28 days after third vaccination up to Day 365 will be summarised by treatment group and by SOC and PT.

#### 17.2. Deaths

If any subjects die during the study, the information will be presented in a data listing.

#### 17.3. Safety Laboratory Evaluations

Clinical laboratory results will be included in the reporting of this study for Haematology, Serum Chemistry and Urinalysis. A list of laboratory assessments to be included in the outputs is included in Appendix 2 of the protocol, Table 6. Presentations will use units, as provided by the labs.

Protocol-specified clinical laboratory tests will be summarized by treatment using descriptive statistics. Clinical laboratory data collected during study conduct, which were not required per protocol, such as for special testing to evaluate an AE, will be listed separately and not summarized.

Quantitative laboratory measurements reported as "< X", i.e. below the lower limit of quantification (BLQ), or "> X", i.e. above the upper limit of quantification (ULQ), will be converted to X for the purpose of quantitative summaries, but will be presented as recorded, i.e. as "< X" or "> X" in the listings.

The following summaries will be provided for laboratory data:

- Observed and change from baseline by visit for each treatment (for quantitative measurements)
- Incidence of abnormal values according to normal range criteria
- Listing of lab results outside the normal range

#### 17.3.1. **Laboratory Reference Ranges**

Quantitative laboratory measurements will be compared with the relevant laboratory reference ranges and categorized as:

- Low: Below the lower limit of the laboratory reference range.
- Normal: Within the laboratory reference range (upper and lower limit included).
- High: Above the upper limit of the laboratory reference range.

\\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\BIOS\MinervaX\GBS-Document:

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS TP BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

Clinical laboratory reference/normal ranges will be listed.

#### 17.4. Vital Signs

The following Vital Signs measurements will be reported for this study:

- Resting Systolic and Diastolic Blood Pressure (mmHg) and Pulse Rate (bpm)
- Oral body temperature (°C)

The following summary will be provided for vital signs data:

• Observed and change from baseline by visit for each treatment

# 17.5. Physical Examination

Physical exam dates will be listed only. New abnormalities occurring after administration of study medication that are clinically significant will be recorded as adverse events.

#### 18. DATA NOT SUMMARIZED OR PRESENTED

The other variables and/or domains not summarized or presented are:

Comments

These domains and/or variables will not be summarized or presented, but will be available in the clinical study database, SDTM and/or ADaM datasets.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\\BIOS\\MinervaX\\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

#### APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS

#### **Dates & Times**

Depending on data available, dates and times will take the form yyyy-mm-ddThh:mm:ss.

# **Spelling Format**

English UK

# **Presentation of Treatment Groups**

For outputs, treatment groups will be represented as follows and in the given order:

| Treatment Group | For Tables and Figures | For Listings (include if different to tables) |
|---|---|---|
| Healthy Older Adult GBS-NN/NN2 50 µg | HOA GBS-NN/NN2 50 μg | |
| Healthy Older Adult GBS-<br>NN/NN2 125 μg | HOA GBS-NN/NN2 125 μg | |
| Healthy Older Adult<br>Placebo | HOA Placebo | |
| Obese and/or Diabetic<br>Older Adult GBS-NN/NN2<br>50 µg | O/DOA GBS-NN/NN2 50 μg | |
| Obese and/or Diabetic<br>Older Adult GBS-NN/NN2<br>125 µg | O/DOA GBS-NN/NN2 125 μg | |
| Obese and/or Diabetic Older Adult Placebo | O/DOA Placebo | |

# Listings

All listings will be ordered by the following (unless otherwise indicated in the template):

- Participating category (healthy old adults vs obese/diabetic old adults), randomized treatment group (or treatment received if it's a safety output), first by active dose [by ascending treatment dose group] and then placebo,
- Center-subject ID,
- Date (where applicable),

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp ops\\BIOS\\MinervaX\\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005



Analysis Plan 

• For listings where non-randomized subjects are included, these will appear in a category after the randomized treatment groups labeled 'Not Randomized'.

Document: \\dccar2dnetvnasc01p-lan1.quintiles.net\cp\_ops\BIOS\MinervaX\GBS-

NN\_NN2\MVX0006\Biostatistics\Documentation\SAP


Template No.: CS\_TP\_BS016 Revision 7 Reference: CS\_WI\_BS005

# Statistical Analysis Plan - V1.0 - SAP or PK-PD Sections Thereof - 23-Apr-2024

# **Electronic Signature Manifestation**

This page is a manifestation of the electronic signature(s) used in compliance with the organization's electronic signature policies and procedures.

| Signer Full<br>Name | Meaning of Signature | <b>Date and Time</b> |
|---|---|---|
| | Document Approval (I certify that I have the education, training and experience to perform this task) | 23 Apr 2024<br>08:45:14 UTC |
| | Document Approval (I certify that I have the education, training and experience to perform this task) | 23 Apr 2024<br>08:49:09 UTC |